CLINICAL TRIAL: NCT00126750
Title: MI-Plus: Web-enhanced Guideline Implementation for Post MI CBOC Patients
Brief Title: Web-Enhanced Guideline Implementation for Post MI CBOC Patients
Acronym: VA MI Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SDR 03-090
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Myocardial Infarction; Comorbidity
Keywords: Myocardial Infarction; Comorbidities; Guidelines; Computer Assisted Instruction; Physician Practice Instruction; Online Systems
MeSH Terms: conditions — Myocardial Infarction | interventions — Drug Interactions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: VA MI Plus Interactive

INTERVENTIONS:
Behavioral: VA MI Plus Interactive — The experimental intervention, customized to the individual clinician in real-time consists of Internet learning modules integrating case-based education with audit, feedback, and benchmarking of practice profiles.

SUMMARY:
To assist busy primary care clinicians in VA Community Based Outpatient Clinics (CBOCs) in managing complex patients by providing a single, interactive, and personalized source of information regarding applicable guidelines for post-MI patients. Specifically, 1) the investigators will identify barriers to provider adherence to guidelines within VHA clinics; 2) Apply guideline-based performance measures to electronic medical records (CPRS) and associated administrative data; 3) Implement the interactive Internet intervention developed by the NHLBI study, after inclusion of VA-specific components, including performance feedback for CBOC clinicians; and 4) Test hypotheses on the intervention's effectiveness, sustainability, and cost-effectiveness in both the VA and Medicare populations. This will include a randomized controlled trial with the CBOC as a unit of randomization.

DETAILED DESCRIPTION:
Some 7.1 million Americans and an estimated 250,000 Veterans actively using VHA are Myocardial Infarction (MI) survivors. To date, most guideline interventions focus on a single patient condition, but ambulatory post-MI patients are frequently more complex, multiple comorbidities, and conflicting guidelines applicable to them. For example, whereas JNC-6 guidelines for the treatment of hypertension suggest pharmacological treatment at blood pressures above 140/80 mm Hg, to be initiated with diuretics or beta-blockers as first line agents, other guidance suggests that for post-MI patients with diabetes, treatment cut-offs should be lower and ACE-inhibitors may be considered as optimal first-line agents. On October 1, 2002, the University of Alabama at Birmingham (UAB) began a study funded by the National Heart, Lung, and Blood institute (NHLBI) as an RO1 (Kiefe, PI (25%), Weissman, co-PI (20%)) to conduct a randomized trial, MI-plus to increase provider adherence to guidelines for post-MI patients. That NHLBI-funded study targets Medicare beneficiaries and their primary care providers in Alabama. Its primary goal is to develop and test with a randomized controlled trial, an Internet-based multimodal guideline implementation strategy. The investigators propose, herewith, to extend and adapt this study to a nationwide sample of VA post-MI patients and their primary care providers in the VA.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects are defined as any VA-employed physician, PA, or CRNP who is a CBOC provider. All such providers will be offered the opportunity to participate and will have the option to agree to participate or not. Performance measure data from records of post-MI patients of the above providers will be extracted to test the experimental intervention. (Note: No individually identifying patient information will be extracted.) All VA-employed CBOC providers (physicians, PAs, CRNPs) will be offered the opportunity to participate in this study. Any subject may refuse to participate or to discontinue participation at will at any point in the study without consequence.

Exclusion Criteria:

Potential subjects must be VA-employed physician, PA, or CRNP who is a CBOC provider. No such healthcare providers will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 847 (Actual)
Dates: Start 2003-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Houston, MD MPH, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford; Ellen Funkhouser, DrPH MS BS, Principal Investigator — VA Medical Center, Birmingham
Locations (41):
- United States (40):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Fayetteville, AR, Fayetteville, Arkansas
  - Long Beach, Long Beach, California
  - VA Medical Center, San Francisco, California
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - VA Medical Center, Miami, Miami, Florida
  - VA Medical Center, Decatur, Decatur, Georgia
  - Jesse Brown VAMC (WestSide Division), Chicago, Illinois
  - VA Illiana Health Care System, Danville, Illinois
  - VA Medical Center Iowa City, Iowa City, Iowa
  - VA Eastern Kansas Health Care System - Topeka, Topeka, Kansas
  - Robert J. Dole VAMC & ROC, Wichita, Kansas
  - VA Medical Center, Louisville, Louisville, Kentucky
  - Overton Brooks VA Medical Center, Shreveport, LA, Shreveport, Louisiana
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, Massachusetts
  - VA Boston Health Care System, Jamaica Plain, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Battle Creek, MI, Battle Creek, Michigan
  - VA Gulf Coast Veterans Health Care System, Biloxi, Mississippi
  - Harry S. Truman Memorial VA Medical Center, Columbia, Missouri
  - Kansas City VA Medical Center, Kansas City, Missouri
  - VA Medical Center, St Louis, St Louis, Missouri
  - VA New Jersey Health Care System, East Orange, East Orange, New Jersey
  - Albany VA Medical Center: Samuel S. Stratton, Albany, New York
  - No Longer Valid, Use 528A8, Albany, New York
  - Franklin Delano Roosevelt Campus of VAHVHCS, Montrose, New York
  - New York, NY, New York, New York
  - VA Medical Center, Cincinnati, Cincinnati, Ohio
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - Coatesville, PA, Coatesville, Pennsylvania
  - Lebanon, PA, Lebanon, Pennsylvania
  - VA Medical Center, Providence, Providence, Rhode Island
  - Ralph H Johnson VA Medical Center, Charleston, Charleston, South Carolina
  - VA Medical Center, Nashville, Tennessee
  - VA Salt Lake City Health Care System, Salt Lake City, Salt Lake City, Utah
  - VA Medical & Regional Office Center, White River, White River Junction, Vermont
  - William S. Middleton Memorial Veterans Hospital, Madison, Wisconsin
  - Clement J. Zablocki VAMC, Milwaukee, Wisconsin
- San Juan VAMC, San Juan, Puerto Rico

REFERENCES:
- [Result] Funkhouser E, Houston TK, Levine DA, Richman J, Allison JJ, Kiefe CI. Physician and patient influences on provider performance: beta-blockers in postmyocardial infarction management in the MI-Plus study. Circ Cardiovasc Qual Outcomes. 2011 Jan 1;4(1):99-106. doi: 10.1161/CIRCOUTCOMES.110.942318. Epub 2010 Dec 7. PMID 21139090
- [Result] Schoen MJ, Tipton EF, Houston TK, Funkhouser E, Levine DA, Estrada CA, Allison JJ, Williams OD, Kiefe CI. Characteristics that predict physician participation in a Web-based CME activity: the MI-Plus study. J Contin Educ Health Prof. 2009 Fall;29(4):246-53. doi: 10.1002/chp.20043. PMID 19998447
- [Result] Levine DA, Funkhouser EM, Houston TK, Gerald JK, Johnson-Roe N, Allison JJ, Richman J, Kiefe CI. Improving care after myocardial infarction using a 2-year internet-delivered intervention: the Department of Veterans Affairs myocardial infarction-plus cluster-randomized trial. Arch Intern Med. 2011 Nov 28;171(21):1910-7. doi: 10.1001/archinternmed.2011.498. PMID 22123798
- [Result] Funkhouser E, Levine DA, Gerald JK, Houston TK, Johnson NK, Allison JJ, Kiefe CI. Recruitment activities for a nationwide, population-based, group-randomized trial: the VA MI-Plus study. Implement Sci. 2011 Sep 9;6:105. doi: 10.1186/1748-5908-6-105. PMID 21906278
- [Result] Ahern DK, Woods SS, Lightowler MC, Finley SW, Houston TK. Promise of and potential for patient-facing technologies to enable meaningful use. Am J Prev Med. 2011 May;40(5 Suppl 2):S162-72. doi: 10.1016/j.amepre.2011.01.005. PMID 21521591
- [Result] Houston TK, Funkhouser E, Allison JJ, Levine DA, Williams OD, Kiefe CI. Multiple measures of provider participation in Internet delivered interventions. Stud Health Technol Inform. 2007;129(Pt 2):1401-5. PMID 17911944
- [Result] Bloch MJ, Basile JN. Analysis of Recent Papers in Hypertension. J Clin Hypertens (Greenwich). 2009 May;11(5):292-95. doi: 10.1111/j.1751-7176.2009.00115.x. No abstract available. PMID 19534038
- [Result] Basile J. Shifting paradigms in defining and treating hypertension: addressing global risk with combination therapy. J Clin Hypertens (Greenwich). 2008 Jan;10(1 Suppl 1):2-3. doi: 10.1111/j.1524-6175.2007.08026.x. No abstract available. PMID 18174777
- [Result] Basile J. The importance of prompt blood pressure control. J Clin Hypertens (Greenwich). 2008 Jan;10(1 Suppl 1):13-9. doi: 10.1111/j.1524-6175.2007.08027.x. PMID 18174779
- [Result] Jamerson KA, Basile J. Prompt, aggressive BP lowering in high-risk patients. J Clin Hypertens (Greenwich). 2008 Jan;10(1 Suppl 1):40-8. doi: 10.1111/j.1524-6175.2007.08145.x. PMID 18174783
- [Result] Cushman WC, Ford CE, Einhorn PT, Wright JT Jr, Preston RA, Davis BR, Basile JN, Whelton PK, Weiss RJ, Bastien A, Courtney DL, Hamilton BP, Kirchner K, Louis GT, Retta TM, Vidt DG; ALLHAT Collaborative Research Group. Blood pressure control by drug group in the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). J Clin Hypertens (Greenwich). 2008 Oct;10(10):751-60. doi: 10.1111/j.1751-7176.2008.00015.x. PMID 19090876
- [Result] Yu FB, Menachemi N, Berner ES, Allison JJ, Weissman NW, Houston TK. Full implementation of computerized physician order entry and medication-related quality outcomes: a study of 3364 hospitals. Am J Med Qual. 2009 Jul-Aug;24(4):278-86. doi: 10.1177/1062860609333626. Epub 2009 Jun 5. PMID 19502568
- [Result] Levine DA, Allison JJ, Cherrington A, Richman J, Scarinci IC, Houston TK. Disparities in self-monitoring of blood glucose among low-income ethnic minority populations with diabetes, United States. Ethn Dis. 2009 Spring;19(2):97-103. PMID 19537217
- [Result] Houston TK, Richman JS, Ray MN, Allison JJ, Gilbert GH, Shewchuk RM, Kohler CL, Kiefe CI; DPBRN Collaborative Group. Internet delivered support for tobacco control in dental practice: randomized controlled trial. J Med Internet Res. 2008 Nov 4;10(5):e38. doi: 10.2196/jmir.1095. PMID 18984559
- [Result] Miller MJ, Allison JJ, Schmitt MR, Ray MN, Funkhouser EM, Cobaugh DJ, Saag KG, LaCivita C. Using single-item health literacy screening questions to identify patients who read written nonsteroidal anti-inflammatory medicine information provided at pharmacies. J Health Commun. 2010 Jun;15(4):413-27. doi: 10.1080/10810731003753091. PMID 20574879

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Among 66 eligible medical centers, the investigators recruited 48 affiliated with 219 clinics, including 957 providers in 26 states, the VIrgin Islands, and Puerto Rico; of these, 168 clinics were randomized (ie, had >1 provider enroll)
Pre-assignment Details: Clinics were randomized when first eligible provider at that clinic logged on to the Web site.
Groups:
- Intervention Group: The intervention included a multicomponent Web site and pushed e-mail cues with educational content.
- Control Group: Providers in control clinics were sent a link to an existing VA Web site that contained links to a wide range of clinical guidelines for various medical conditions.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 385 (Number of providers from 84 clinics) | 462 (Number of providers from 84 clinics)
Completed | 205 (Total providers at participating clinic locations were given the option to 'enroll'.) | 196 (Total providers at clinic locations were given the option to 'enroll'.)
Not Completed | 180 | 266

BASELINE CHARACTERISTICS:
Groups:
- Intervention Arm/Group: Providers from eligible clinics that were allocated to the intervention arm.
- Control Arm/Group: Providers from eligible clinics that were allocated to the control arm.
- Total: Total of all reporting groups
Arm/Group | Intervention Arm/Group | Control Arm/Group | Total
Number analyzed (Participants) | 385 | 462 | 847
Age, Categorical [Number] — Age data not collected
  value
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number] — Gender data not collected
  value
    Gender | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Was the Performance of Each Provider on Each of Seven Clinical Indicators
Description: The investigators used an intent-to-treat approach for our main analysis, basing our outcome measures on provider's eligible patient population in each of the clinics. Performance improvement was calculated at the change (before vs after the intervention) the percentage of provider's patients with each clinical indicator. 1) change in the percentage of patients with improvements in LDL. Improvement defined as LDL-C level < previous 18 mos; 2) Change in the percentage of patients with improvements in A1c. Improvement defined as HbA1c level < previous 18 mos; 3) Change in percentage of patients prescribed Beta Blockers; 4) Change in the percentage of patients prescribed Statins; 5) Change in the percentage of patients prescribed ACEI or ARB; 6) Change in percentage of patients reaching target goal for LDL-C (<100mg/dL); 7) Change in percentage of patients reaching target goal for HbA1c (<8%).
Time Frame: 1/1/02 - 12/31/08
Measure: Number; unit: percentage of provider's patients
Groups:
- Intervention: Intervention Providers received an interactive, educational website and motivational reminders.
- Control: Control Providers received a link to VA practice guidelines.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 385 | 462
percentage of provider's patients
  Change in % of patients w/ improvement in LDL | 2.8 | 2.1
  Change in % of patients w/ improvement in HbA1c | 11.5 | 9.5
  Change in % of patients prescribed B-Blockers | 15.5 | 12.1
  Change in % patients prescribed Statins | 8.5 | 7.5
  Change in % of patients prescribed ACEI or ARB | 4.9 | 2.9
  Change in % of patients reaching target LDL | 19.9 | 15.2
  Change in % of patients reaching target HbA1c | 6 | .7

ADVERSE EVENTS:
Groups:
- Intervention Group; Control Group: Because this was an RCT of clinics and providers utilization of web-based intervention, no serious (or non-serious) adverse events were collected.
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes